CLINICAL TRIAL: NCT01158690
Title: Intimate Partner Violence and Pregnancy, a Randomised Controlled Trial on the Effect of a Resource Card on the Incidence of Intimate Partner Violence
Brief Title: Intimate Partner Violence and Pregnancy, a Perinatal Care Intervention Study
Acronym: MOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); International Centre for Reproductive Health, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2010/093
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Intimate Partner Violence
Keywords: Intimate partner violence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- resource card group (Experimental): The intervention group will receive an envelope with a gift voucher and a resource card (wallet size card with on the one side safety measures and on the other side contact details of resources for violence).
  Interventions: Other: resource card
- control group (Active Comparator): The control group will receive the same envelop with a gift voucher and a letter of thanks.
  Interventions: Other: no resource card

INTERVENTIONS:
Other: resource card — the intervention group receives an envelop with resource card
  Arms: resource card group
Other: no resource card — the control group receives an envelop without resource card
  Arms: control group

SUMMARY:
The study composes of two large parts, in particular a large scale prevalence/incidence study and a single-blind randomised controlled trial (RCT). The prevalence/incidence study aims to determine the prevalence/incidence of physical, psychological and sexual violence in a pregnant population. The study population is recruited through the prenatal consultation of more or less 15 hospitals in Belgium. The respondents fill out a questionnaire on the spot minimum one time during pregnancy. Based on this questionnaire, the investigators aim to recruit 150 victims of intimate partner violence (IPV) to participate in the second part of the study. The RCT aims to evaluate if there is a safe and effective way to reduce IPV within the perinatal care setting. The investigators hypothesise that screening pregnant women for violence in combination with handing out a resource card, has the potential of interrupting the IPV and increase help-seeking behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Dutch-, French- or English speaking
* Victim of intimate partner violence based on the questionnaire
* Accessible through telephone and no safety problems

Exclusion Criteria:

* Not Dutch-, French- or English speaking
* Not a victim of intimate partner violence one year before or during pregnancy
* Not accessible through telephone and/or safety problems

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Impact of the resource card on the evolution of the partner violence within a sample of pregnant victims of partner violence | 6 months after receipt of the resource card
Impact of the resource card on the evolution of the partner violence within a sample of pregnant victims of partner violence | 12 months after the receipt of the resource card

SECONDARY OUTCOMES:
Impact of a resource card on the evolution of the help-seeking behaviour | 6 months after receipt of the resource card
Impact of a resource card on the evolution of the help-seeking behaviour | 12 months after receipt of the resource card

CONTACTS AND LOCATIONS:
Overall Officials: Marleen Temmerman, MD, PhD, Principal Investigator — University Ghent
Locations (12):
- Belgium (12):
  - OLV Ziekenhuis Aalst, Aalst
  - UZA, Antwerp
  - ZNA Middelheim Antwerpen, Antwerp
  - AZ Sint-Jan Brugge, Bruges
  - AZ Monica Deurne, Deurne
  - ZOL Genk, Genk
  - AZ Jan Palfijn Gent, Ghent
  - Ghent University Hospital, Ghent
  - Virga Jesse Hasselt, Hasselt
  - AZ Groeninge Kortrijk, Kortrijk
  - OLV van Lourdes ziekenhuis Waregem, Waregem
  - AZ Sint-Augustinus Ziekenhuis Wilrijk, Wilrijk

REFERENCES:
- [Derived] Van Parys AS, Deschepper E, Roelens K, Temmerman M, Verstraelen H. The impact of a referral card-based intervention on intimate partner violence, psychosocial health, help-seeking and safety behaviour during pregnancy and postpartum: a randomized controlled trial. BMC Pregnancy Childbirth. 2017 Oct 6;17(1):346. doi: 10.1186/s12884-017-1519-x. PMID 28985722